CLINICAL TRIAL: NCT03686527
Title: Myocardial Function of the Setonis Aortic Valve Before and Beyond Valve
Brief Title: Myocardial Function of the Setonis Aortic Valve Before and Beyond Valve Replacement
Acronym: AOMYOC
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC12_8974 AOMYOC
Record Dates: First submitted 2018-09-25; First posted 2018-09-27 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2018-09

CONDITIONS: Myocardial Function of the Stenosis Aortic Valve Before and Beyond Valve Replacement

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Echocardiography
  Interventions: Procedure: stenosis aortic valve
- MRI Fibrosis
  Interventions: Procedure: stenosis aortic valve

INTERVENTIONS:
Procedure: stenosis aortic valve — The exams to be realized :
  * a clinical examination with blood pressure
  * a 12-lead surface electrocardiogram
  * a standard biological assessment including NTproBNP (Brain Natriuretic Peptide)
  * Transthoracic echocardiography at baseline and 12 months after the aortic valve intervention on the (according to recommendations)
  * a cardiac MRI looking for fibrosis myocardial

SUMMARY:
Study the consequences on heart muscle of the stenosis aortic valve before and after the replacement procedure, the repercussion on heart. Study the impact on the heart of "sick" valve can affect on "well-being" and prognosis in the year following the surgery.

ELIGIBILITY:
Inclusion Criteria:

* major patient freely accepting to participate in the study
* non-opposition signed
* aortic surface <1cm² or <0.6cm² / m² of indication surgical restraint
* oriented to short interventional management surgical term
* LVEF Left ventricular ejection fraction> 50%
* In the subgroup "MRI-fibrosis", absence of indication for performing MRI

Exclusion Criteria:

* patient under guardianship, curatorship or safeguard of justice
* minor patient
* pregnant woman
* patient with significant polyvalvulopathy for which it is from the start programmed more than aortic valve replacement
* patient with severe coronary artery disease requiring revascularization
* allergy to the contrast product

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with tight aortic stenosis with an indication of surgical treatment.
Sampling Method: Non-Probability Sample
Enrollment: 277 (Actual)
Dates: Start 2018-01-11 (Actual); Primary Completion 2019-01-11 (Actual); Study Completion 2019-01-11 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is a composite endpoint: all-cause death, cardiovascular hospitalization: cardiac decompensation, atrial fibrillation within 12 months of surgical or percutaneous aortic valve replacement. | 1 day of inclusion

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Rennes, Rennes, Brittany Region, France